CLINICAL TRIAL: NCT05412108
Title: Prospective Evaluation of Complications of MidLine Catheters in the ICU
Acronym: COMIDREA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2020/S03/13
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Catheter Complications
Keywords: Midline catheter; ICU Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Midline catheters (MCs) are peripheral catheters inserted into a vein in the arm above the elbow crease, with the tip in the axillary vein. As such, they do not enter the central venous circulation and are therefore not considered central venous catheters.

The main complications associated with CM are accidental removal, leakage, subcutaneous diffusion and occlusion. Severe complications include deep vein thrombosis (DVT) and catheter-related bacteremia (CRB). There is very little data on the use of CMs in intensive care units (ICU).

Resuscitation patients are more likely to develop severe catheter-related complications such as deep vein thrombosis and catheter-related infections. While the use of CMs in patients appears to be associated with a low risk of complications, this may not be the case in resuscitation patients.

Investigator therefore proposes to conduct a prospective observational study to determine the frequency and type of complications associated with CMs when they are implanted and used in ICU. In addition, investigator will attempt to determine whether risk factors predictive of complications can be identified. In addition, this study will evaluate whether the use of CMs can reduce the duration of central venous catheter maintenance in the ICU and the risk of central venous catheter-related infections.

ELIGIBILITY:
Inclusion Criteria:

* ICU Hospitalization
* Indication for MidLine catheter placement during the stay

Exclusion Criteria:

* Minor or protected adult
* Pregnant woman
* Local contraindication to the placement of a CM

  * Local infection
  * Venous thrombosis
  * Existing arteriovenous fistula or vascular network to be protected for a fistula for chronic dialysis
  * Paralysis of the limb
* Need for administration of contraindicated solutions on the peripheral venous route:

  * Catecholamines: Noradrenaline, adrenaline (dose greater than 0.2µg/kg/min)
  * Total parenteral nutrition
  * Glucose solutions at a concentration >20
  * Potassium at a concentration >0.1mEq/ml
  * Vesicants
  * Fluids with pH <5 or >9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU for whom an indication for placement of a MidLine catheter is identified during their ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Describe the incidence of severe complications associated with the use of CMs in ICUs | From midline catheter placement to hospital discharge (up to 28 days)
  The severe complications identified will be symptomatic deep vein thrombosis, symptomatic pulmonary embolism, catheter-related infections

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France